CLINICAL TRIAL: NCT03191396
Title: Efficacy and Safety of Semaglutide 1.0 mg Once-weekly Versus Liraglutide 1.2 mg Once-daily as add-on to 1-3 Oral Anti-diabetic Drugs (OADs) in Subjects With Type 2 Diabetes
Brief Title: Research Study Comparing a New Medicine Semaglutide to Liraglutide in People With Type 2 Diabetes
Acronym: SUSTAIN 10
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9535-4339; 2016-004965-22 (Registry Identifier: EudraCT); U1111-1190-5868 (Other: World Health Organization (WHO))
Record Dates: First submitted 2017-06-16; First posted 2017-06-19 (Actual); Results first posted 2019-08-28 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide; Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Semaglutide (Experimental): Half the study participants are randomised to receive semaglutide
  Interventions: Drug: Semaglutide
- Liraglutide (Active Comparator): Half the study participants are randomised to receive liraglutide
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Semaglutide — Dose gradually increased to 1.0 mg, given s.c. (under the skin), once-weekly for 30 weeks. Participants will remain on their pre-study anti-diabetic drugs (tablets), if any
  Arms: Semaglutide
Drug: Liraglutide — Dose gradually increased to 1.2 mg, given s.c. once-daily for 30 weeks. Participants will remain on their pre-study anti-diabetic drugs, if any
  Arms: Liraglutide

SUMMARY:
This study is conducted in Europe. The aim of the study is to compare the effect of semaglutide subcutaneous (s.c., under the skin) 1.0 mg once-weekly to liraglutide s.c.1.2 mg once-daily on blood sugar levels after 30 weeks of treatment in people with type 2 diabetes. The study will last approximately 9 months (37 weeks). Each participant will have 7 visits at the clinic and 3 phone calls with the study doctor. At the visits, participants will have a number of tests, for example: general health checks, blood samples, heart and eye checks etc. Participants will also fill in some forms about their health and satisfaction with their diabetes treatment.

ELIGIBILITY:
Inclusion Criteria: - Male or female, age 18 years or older at the time of signing informed consent - Diagnosed with type 2 diabetes mellitus - HbA1c of 7.0-11.0 % (53 - 97 mmol/mol) (both inclusive) - Stable daily dose(s) including any of the following anti-diabetic drug(s) or combination regimens 90 days prior to the day of screening: a) Biguanides (metformin above or equal to 1500 mg or maximum tolerated dose documented in the subject's medical record). b) Sulphonylureas (above or equal to half of the maximum approved dose according to local label or maximum tolerated dose as documented in subject medical record). c) SGLT-2 inhibitors (above or equal to half of the maximum approved dose according to local label or maximum tolerated dose as documented in subject medical record) Exclusion Criteria: - Family or personal history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma. Family is defined as a first degree relative - History or presence of pancreatitis (acute or chronic) - History of diabetic ketoacidosis - Any of the following: myocardial infarction, stroke, hospitalization for unstable angina or transient ischaemic attack within the past 180 days prior to the day of screening - Subjects presently classified as being in New York Heart Association (NYHA) Class IV - Planned coronary, carotid or peripheral artery revascularisation known on the day of screening - Renal impairment measured as estimated Glomerular Filtration Rate (eGFR) value of below 30 ml/min/1.73 sqm as defined by KDIGO 2012 classification - Impaired liver function, defined as ALT above or equal to 2.5 times upper normal limit at screening - Proliferative retinopathy or maculopathy requiring acute treatment. Verified by fundus photography or dilated fundoscopy performed within the past 90 days prior to randomisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 577 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2018-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (86):
- Bulgaria (9):
  - Novo Nordisk Investigational Site, Burgas
  - Novo Nordisk Investigational Site, Dupnitsa
  - Novo Nordisk Investigational Site, Lukovit
  - Novo Nordisk Investigational Site, Madan
  - Novo Nordisk Investigational Site, Petrich
  - Novo Nordisk Investigational Site, Rousse
  - Novo Nordisk Investigational Site, Sliven
  - Novo Nordisk Investigational Site, Sofia
  - Novo Nordisk Investigational Site, Vratsa
- Czechia (3):
  - Novo Nordisk Investigational Site, Brno
  - Novo Nordisk Investigational Site, Náchod
  - Novo Nordisk Investigational Site, Prague
- Finland (8):
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Jyväskylä
  - Novo Nordisk Investigational Site, Kuusamo
  - Novo Nordisk Investigational Site, Lahti
  - Novo Nordisk Investigational Site, Oulu
  - Novo Nordisk Investigational Site, Rauma
  - Novo Nordisk Investigational Site, Turku
  - Novo Nordisk Investigational Site, Varkaus
- France (14):
  - Novo Nordisk Investigational Site, Béziers
  - Novo Nordisk Investigational Site, Dambach-la-Ville
  - Novo Nordisk Investigational Site, Dijon
  - Novo Nordisk Investigational Site, La Rochelle
  - Novo Nordisk Investigational Site, Le Coudray
  - Novo Nordisk Investigational Site, Le Creusot
  - Novo Nordisk Investigational Site, Nantes
  - Novo Nordisk Investigational Site, Obernai
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Perpignan
  - Novo Nordisk Investigational Site, Schiltigheim
  - Novo Nordisk Investigational Site, Strasbourg
  - Novo Nordisk Investigational Site, Vandœuvre-lès-Nancy
  - Novo Nordisk Investigational Site, Vénissieux
- Germany (6):
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Essen
  - Novo Nordisk Investigational Site, Falkensee
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Saint Ingbert-Oberwürzbach
  - Novo Nordisk Investigational Site, Stuttgart
- Hungary (7):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Nagykanizsa
  - Novo Nordisk Investigational Site, Pécs
  - Novo Nordisk Investigational Site, Siófok
  - Novo Nordisk Investigational Site, Szolnok
  - Novo Nordisk Investigational Site, Tatabánya
  - Novo Nordisk Investigational Site, Zalaegerszeg
- Italy (5):
  - Novo Nordisk Investigational Site, Bergamo
  - Novo Nordisk Investigational Site, Como
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Pavia
  - Novo Nordisk Investigational Site, Rome
- Poland (2):
  - Novo Nordisk Investigational Site, Lublin
  - Novo Nordisk Investigational Site, Szczecin
- Slovenia (4):
  - Novo Nordisk Investigational Site, Celje
  - Novo Nordisk Investigational Site, Jesenice
  - Novo Nordisk Investigational Site, Koper
  - Novo Nordisk Investigational Site, Ljubljana
- Spain (6):
  - Novo Nordisk Investigational Site, Alcorcón
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, La Roca Del Vallés
  - Novo Nordisk Investigational Site, Palma de Mallorca
  - Novo Nordisk Investigational Site, Valladolid
  - Novo Nordisk Investigational Site, Vic (Barcelona)
- Sweden (5):
  - Novo Nordisk Investigational Site, Ängelholm
  - Novo Nordisk Investigational Site, Kristianstad
  - Novo Nordisk Investigational Site, Lund
  - Novo Nordisk Investigational Site, Örebro
  - Novo Nordisk Investigational Site, Stockholm
- United Kingdom (17):
  - Novo Nordisk Investigational Site, Blackpool
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Coventry
  - Novo Nordisk Investigational Site, Crewe
  - Novo Nordisk Investigational Site, Faringdon
  - Novo Nordisk Investigational Site, Hinckley
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Northwood
  - Novo Nordisk Investigational Site, Norwich
  - Novo Nordisk Investigational Site, Nuneaton
  - Novo Nordisk Investigational Site, Rhyl
  - Novo Nordisk Investigational Site, Rotherham
  - Novo Nordisk Investigational Site, Sidcup
  - Novo Nordisk Investigational Site, Southampton
  - Novo Nordisk Investigational Site, St Helens
  - Novo Nordisk Investigational Site, Truro
  - Novo Nordisk Investigational Site, Watford

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Result] Capehorn MS, Catarig AM, Furberg JK, Janez A, Price HC, Tadayon S, Verges B, Marre M. Efficacy and safety of once-weekly semaglutide 1.0mg vs once-daily liraglutide 1.2mg as add-on to 1-3 oral antidiabetic drugs in subjects with type 2 diabetes (SUSTAIN 10). Diabetes Metab. 2020 Apr;46(2):100-109. doi: 10.1016/j.diabet.2019.101117. Epub 2019 Sep 17. PMID 31539622
- [Derived] Capehorn M, Ghani Y, Hindsberger C, Johansen P, Jodar E. Once-Weekly Semaglutide Reduces HbA1c and Body Weight in Patients with Type 2 Diabetes Regardless of Background Common OAD: a Subgroup Analysis from SUSTAIN 2-4 and 10. Diabetes Ther. 2020 May;11(5):1061-1075. doi: 10.1007/s13300-020-00796-z. Epub 2020 Mar 19. PMID 32193837

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 77 sites in 11 countries as follows (number of sites that screened subjects/ number of sites that randomised subjects):
  Bulgaria (9/ 9); Czech Republic (5/ 5); Finland (8/ 8); France (8/ 8); Hungary (8/ 8); Italy (4/ 4); Poland (3/ 3); Slovenia (4/ 4); Spain (5/ 5); Sweden (6/ 6); United Kingdom (17/ 17)
Pre-assignment Details: After screening, subjects were required to continue their oral anti-diabetic drug (OAD) pre-trial background medication (i.e. metformin, Sodium-glucose co-transporter-2 (SGLT-2) inhibitors, sulphonyl ureas, or combinations of these) throughout the entire trial.
Groups:
- Semaglutide 1.0 mg: Subjects received 1.0 mg semaglutide once-weekly for 30 weeks (including 8-week dose escalation period). Semaglutide was administered subcutaneously by injections in the thigh, abdomen or upper arm once weekly on the same weekday. Subjects started semaglutide at 0.25 mg and were dose escalated in 4-week increments until the final maintenance dose of 1.0 mg was reached (i.e. 0.25 mg from week 0 to week 4, 0.5 mg from week 4 to week 8 and 1.0 mg from week 8 to week 30). Subjects also continued their OAD pre-trial background medication (i.e. metformin, SGLT-2 inhibitors, sulphonyl ureas, or combinations of these).
- Liraglutide 1.2 mg: Subjects received 1.2 mg liraglutide once-daily for 30 weeks (including 1-week dose escalation period). Liraglutide was administered subcutaneously by injections in the thigh, abdomen or upper arm once-daily and the time of injection was to be consistent from one day to another. Subjects started liraglutide at 0.6 mg for 1 week and then were dose escalated to the maintenance dose of 1.2 mg. Subjects also continued their OAD pre-trial background medication (i.e. metformin, SGLT-2 inhibitors, sulphonyl ureas, or combinations of these).
Period: Overall Study
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Started | 290 | 287
Completed | 287 | 282
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 0 | 3
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg | Total
Number analyzed (Participants) | 290 | 287 | 577
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.1 (10.5) | 58.9 (10.0) | 59.5 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 120 | 250
  Male | 160 | 167 | 327
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 268 | 269 | 537
  Unknown or Not Reported | 16 | 15 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 264 | 268 | 532
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c
Description: Mean change from baseline (week 0) to week 30 in glycosylated haemoglobin (HbA1c) %. The endpoint was evaluated based on the 'on-treatment without rescue medication period' where subjects were considered treated with trial product, but had not yet initiated rescue medication. Missing data were imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates.
Time Frame: Week 0, week 30
Population: Full analysis set (FAS), which included all randomised participants.
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated haemoglobin
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 290 | 287
Percentage of glycosylated haemoglobin | -1.7 (0.9) | -1.1 (1.0)
Statistical Analysis 1: Comparison: Semaglutide 1.0 mg vs Liraglutide 1.2 mg; The responses are analysed using an ANCOVA with treatment and stratification factor as fixed factors and baseline value as covariate. Before analysis, missing data were multiple imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates; Test type: Non-Inferiority — HbA1c non-inferiority was tested using a non-inferiority margin of 0.3; p < 0.0001, ANCOVA — The non-inferiority p-value is calculated as two times the one-sided p-value from a t-distributed test statistic comparing the treatment contrast with 0.3; Treatment difference = -0.69, 95% CI 2-sided [-0.82 to -0.56] — Semaglutide 1.0 mg - Liraglutide 1.2 mg
Statistical Analysis 2: Comparison: Semaglutide 1.0 mg vs Liraglutide 1.2 mg; Test type: Superiority; p < 0.0001, ANCOVA; Treatment difference = -0.69, 95% CI 2-sided [-0.82 to -0.56] — Semaglutide 1.0 mg - Liraglutide 1.2 mg

2. Secondary Outcome: Change in Body Weight (kg)
Description: Mean change from baseline (week 0) to week 30 in body weight measured in kilograms. Results are based on the 'on-treatment without rescue medication' observation period. Missing data were imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates.
Time Frame: Week 0, week 30
Population: Full analysis set (FAS), which included all randomised participants.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 290 | 287
kg | -5.8 (4.7) | -2.0 (4.1)
Statistical Analysis 1: Comparison: Semaglutide 1.0 mg vs Liraglutide 1.2 mg; Test type: Superiority; p < 0.0001, ANCOVA; Treatment difference = -3.83, 95% CI 2-sided [-4.57 to -3.09] — Semaglutide 1.0 mg - Liraglutide 1.2 mg

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Mean change from baseline in fasting plasma glucose measured in mmol/L. Results are based on the 'on-treatment without rescue medication' observation period. Missing data were imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates.
Time Frame: Week 0, week 30
Population: Full analysis set (FAS), which included all randomised participants. Number analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 290 | 287
mmol/L | -2.65 (2.19) | -1.46 (2.42)

4. Secondary Outcome: Change in Self-measured Plasma Glucose (SMPG), 7 Point Profile: Mean 7-point Profile
Description: Mean change from baseline in 7-point profile. SMPG was recorded at the following 7 time points: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after dinner and at bedtime. The mean of the 7-point SMPG profile, defined as the area under the profile, was calculated using the trapezoidal method and divided by the measurement time. Results are based on the 'on-treatment without rescue medication' observation period. Missing data were imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates.
Time Frame: Week 0, week 30
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 290 | 287
mmol/L | -3.0 (2.0) | -2.1 (2.3)

5. Secondary Outcome: Change in Self-measured Plasma Glucose (SMPG), 7 Point Profile: Mean Post Prandial Increment (Over All Meals)
Description: Mean post prandial glucose incrememts over all meals. Results are based on the on-treatment without rescue medication period. Missing data were imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates.
Time Frame: Week 0, week 30
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 290 | 287
mmol/L | -1.0 (1.8) | -0.4 (1.9)

6. Secondary Outcome: Change in Fasting Blood Lipids: Total Cholesterol
Description: The change from baseline in total cholesterol (measured in mmol/L) is presented as ratio to baseline. Results are based on the on-treatment without rescue medication period. Missing data were imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates.
Time Frame: Week 0, week 30
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 290 | 287
ratio | 0.96 (16.8) | 0.98 (16.9)

7. Secondary Outcome: Change in Fasting Blood Lipids: Low-density Lipoprotein (LDL)-Cholesterol
Description: The change from baseline in LDL cholesterol is presented as ratio to baseline. Results are based on the on-treatment without rescue medication period. Missing data were imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates.
Time Frame: Week 0, week 30
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 290 | 287
ratio | 0.99 (28.3) | 0.99 (27.2)

8. Secondary Outcome: Change in Fasting Blood Lipids: High-density Lipoprotein (HDL)-Cholesterol
Description: The change from baseline in HDL cholesterol is presented as ratio to baseline. Results are based on the on-treatment without rescue medication period. Missing data were imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates.
Time Frame: Week 0, week 30
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 290 | 287
ratio | 1.01 (14.6) | 0.99 (12.9)

9. Secondary Outcome: Change in Fasting Blood Lipids: Triglycerides
Description: The change from baseline in triglycerides is presented as ratio to baseline. Results are based on the on-treatment without rescue medication period. Missing data were imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates.
Time Frame: Week 0, week 30
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 290 | 287
Ratio | 0.83 (41.5) | 0.91 (39.5)

10. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Mean change from baseline (week 0) to week 30 in BMI. BMI was calculated as 'body weight in kg/(height in meters) x (height in meters)'. Results are based on the on-treatment without rescue medication period. Missing data were imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates.
Time Frame: Week 0, week 30
Population: Full analysis set (FAS), which included all randomised participants.
Measure: Mean (Standard Deviation); unit: kg/sqm
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 290 | 287
kg/sqm | -2.0 (1.6) | -0.7 (1.4)

11. Secondary Outcome: Change in Waist Circumference
Description: Mean change in waist circumference (cm) from baseline (week 0) to week 30. Results are based on the on-treatment without rescue medication period. Missing data were imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates.
Time Frame: Week 0, week 30
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 290 | 287
cm | -5.2 (5.6) | -2.4 (4.6)

12. Secondary Outcome: Change in Systolic Blood Pressure
Description: Change in systolic blood pressure from baseline (week 0) to week 30 . Results are based on the on-treatment without rescue medication period. Missing data were imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates.
Time Frame: Week 0, week 30
Population: Full analysis set (FAS), which included all randomised participants.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 290 | 287
mmHg | -4.3 (13.4) | -3.7 (13.8)

13. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Change in diastolic blood pressure from baseline (week 0) to week 30 . Results are based on the on-treatment without rescue medication period. Missing data were imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates.
Time Frame: Week 0, week 30
Population: Full analysis set (FAS), which included all randomised participants.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 290 | 287
mmHg | -1.5 (8.6) | -1.3 (8.4)

14. Secondary Outcome: Change in Body Weight (%)
Description: Mean relative change from baseline in body weight measured in percentage. Results are based on the 'on-treatment without rescue medication' observation period. Missing data were imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates.
Time Frame: Week 0, week 30
Population: Full analysis set (FAS), which included all randomised participants.
Measure: Mean (Standard Deviation); unit: percentage of body weight
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 290 | 287
percentage of body weight | -6.1 (4.9) | -2.0 (4.2)

15. Secondary Outcome: Subjects Who Achieve HbA1c Below 7.0% (53 mmol/Mol), American Diabetes Association (ADA) Target
Description: Percentage of subjects who achieved HbA1c less than 7.0% (53 mmol/mol) according to American Diabetes Association (ADA) target, after 30 weeks of treatment. Results are based on the on-treatment without rescue medication period. Missing data were imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates.
Time Frame: After 30 weeks of treatment
Population: Full analysis set (FAS), which included all randomised participants.
Measure: Number; unit: percentage of participants
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 290 | 287
percentage of participants | 80.4 | 45.9

16. Secondary Outcome: Subjects Who Achieve HbA1c Below or Equal to 6.5% (48 mmol/Mol), American Association of Clinical Endocrinologists (AACE) Target
Description: Percentage of subjects who achieved HbA1c less than 6.5% (48 mmol/mol) according to AACE target,after 30 weeks of treatment. Results are based on the on-treatment without rescue medication period. Missing data were imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates.
Time Frame: After 30 weeks of treatment
Population: Full analysis set (FAS), which included all randomised participants.
Measure: Number; unit: percentage of participants
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 290 | 287
percentage of participants | 58.5 | 24.8

17. Secondary Outcome: Subjects Who Achieve Weight Loss Above or Equal to 3%
Description: Percentage of subjects who achieved weight loss above or equal to 3% after 30 weeks of treatment. Results are based on the on-treatment without rescue medication period. Missing data were imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates.
Time Frame: After 30 weeks of treatment
Population: Full analysis set (FAS), which included all randomised participants.
Measure: Number; unit: percentage of participants
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 290 | 287
percentage of participants | 72.7 | 33.9

18. Secondary Outcome: Subjects Who Achieve Weight Loss Above or Equal to 5%
Description: Percentage of subjects who achieved weight loss above or equal to 5% after 30 weeks of treatment. Results are based on the on-treatment without rescue medication period. Missing data were imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates.
Time Frame: After 30 weeks of treatment
Population: Full analysis set (FAS), which included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 290 | 287
Percentage of participants | 55.9 | 17.7

19. Secondary Outcome: Subjects Who Achieve Weight Loss Above or Equal to 10%
Description: Percentage of subjects who achieved weight loss above or equal to 10% after 30 weeks of treatment. Results are based on the on-treatment without rescue medication period. Missing data were imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates.
Time Frame: After 30 weeks of treatment
Population: Full analysis set (FAS), which included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 290 | 287
Percentage of participants | 19.1 | 4.4

20. Secondary Outcome: Subjects Who Achieve HbA1c Below 7.0% (53 mmol/Mol) Without Severe or Blood Glucose Confirmed Symptomatic Hypoglycaemia Episodes and no Weight Gain
Description: Percentage of subjects who achieved HbA1c below 7.0% (53 mmol/mol) without severe or blood glucose confirmed symptomatic hypoglycaemia episodes and no weight gain, after 30 weeks of treatment. Results are based on the on-treatment without rescue medication period. Missing data were imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates.
Time Frame: After 30 weeks of treatment
Population: Full analysis set (FAS), which included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 290 | 287
Percentage of participants | 75.6 | 36.8

21. Secondary Outcome: Subjects Who Achieve HbA1c Reduction Above or Equal to 1%
Description: Percentage of subjects who achieved weight loss above or equal to 1% after 30 weeks of treatment. Results are based on the on-treatment without rescue medication period. Missing data were imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates.
Time Frame: After 30 weeks of treatment
Population: Full analysis set (FAS), which included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 290 | 287
Percentage of participants | 82.8 | 48.3

22. Secondary Outcome: Subjects Who Achieve HbA1c Reduction Above or Equal to 1% and Weight Loss Above or Equal to 3%
Description: Percentage of subjects who achieved HbA1c reduction above or equal to 1% and weight loss above or equal to 3% after 30 weeks of treatment. Results are based on the on-treatment without rescue medication period. Missing data were imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates.
Time Frame: After 30 weeks of treatment
Population: Full analysis set (FAS), which included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 290 | 287
Percentage of participants | 62.4 | 20.9

23. Secondary Outcome: Subjects Who Achieve HbA1c Reduction Above or Equal to 1% and Weight Loss Above or Equal to 5%
Description: Percentage of subjects who achieved HbA1c reduction above or equal to 1% and weight loss above or equal to 5% after 30 weeks of treatment. Results are based on the on-treatment without rescue medication period. Missing data were imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates.
Time Frame: After 30 weeks of treatment
Population: Full analysis set (FAS), which included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 290 | 287
Percentage of participants | 49.6 | 11.9

24. Secondary Outcome: Subjects Who Achieve HbA1c Reduction Above or Equal to 1% and Weight Loss Above or Equal to 10%
Description: Percentage of subjects who achieved HbA1c reduction above or equal to 1% and weight loss above or equal to 10% after 30 weeks of treatment. Results are based on the on-treatment without rescue medication period. Missing data were imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates.
Time Frame: After 30 weeks of treatment
Population: Full analysis set (FAS), which included all randomised participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 290 | 287
Percentage of participants | 17.1 | 3.6

25. Secondary Outcome: Change in SF-36v2 Short Form Health Survey. Total Summary Scores (Physical Component and Mental Component) and Scores From the 8 Domains
Description: Short form-36 version 2 (SF-36v2) is a 36-item patient-reported survey of patient health that measures the subject's overall health-related quality of life (HRQoL). The questionnaire measures the individual overall HRQoL on 8 domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional and mental health. Each domain is scored using the sum of the individual item responses and normalised relative to the 2009 US reference population. Overall, the domain scores range from around 0-100 (higher scores indicated a better HRQoL), where the range of possible scores depends on the 2009 US reference population for each domain. The two total summary scores (mental and physical summary components) are calculated through weighted sums of the 8 domain scores. The presented result is the change from baseline (week 0) to week 30 in SF-36v2 scores. A positive change in score indicates an improvement since baseline.
Time Frame: Week 0, week 30
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 290 | 287
scores on a scale
  Physical functioning | 1.8 (5.8) | 1.4 (6.6)
  Role-physical: number analyzed (Participants) | 289 | 287
  Role-physical | 1.4 (7.2) | 0.6 (6.7)
  Bodily pain | 2.2 (9.1) | 1.5 (9.8)
  General health | 2.7 (7.9) | 1.6 (7.7)
  Social functioning | 1.7 (8.7) | 0.9 (7.7)
  Role-emotional: number analyzed (Participants) | 289 | 287
  Role-emotional | 1.2 (8.5) | 1.0 (8.0)
  Vitality | 3.0 (8.0) | 1.1 (8.0)
  Mental health | 1.7 (8.2) | 0.3 (7.2)
  Mental component summary: number analyzed (Participants) | 289 | 287
  Mental component summary | 1.7 (7.9) | 0.5 (7.5)
  Physical component summary: number analyzed (Participants) | 289 | 287
  Physical component summary | 2.1 (6.4) | 1.4 (5.9)

26. Secondary Outcome: Change in Diabetes Treatment Satisfaction Questionnaire (DTSQ). Treatment Satisfaction Summary Score (Sum of 6 of 8 Items) and the 8 Items Separately
Description: The DTSQs questionnaire was used to assess subject's treatment satisfaction. This instrument contains 8 items and measures the treatment for diabetes in terms of convenience, flexibility and general feelings regarding treatment. Q 1 = "satisfaction with current treatment"; Q 2 = "hyperglycemia"; Q 3 = "hypoglycemia"; Q 4 = "flexibility"; Q 5 = "convenience"; Q 6 = "understanding of diabetes"; Q 7 = "recommend treatment to others"; and Q 8 = "willingness to continue". Each item is rated on a 7-point Likert scale with a score ranging from 0 (ie, very dissatisfied) to 6 (ie, very satisfied). DTSQ items 2 and 3 are rated differently: 0 reflects 'never' and 6 reflects 'most of the time'. The 'treatment satisfaction' score is the sum of 6 of the 8 DTSQs components (Q 1, 4, 5, 6, 7 and 8) (range 0-36). Higher scores on the DTSQ total score indicate higher treatment satisfaction. The results presented is the change from baseline (week 0) to week 30 in DTSQ scores.
Time Frame: Week 0, week 30
Population: Full analysis set (FAS), which included all randomised participants. Missing data were imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 290 | 287
scores on a scale
  Q1. Satisfaction with current treatment: number analyzed (Participants) | 290 | 286
  Q1. Satisfaction with current treatment | 0.9 (1.7) | 0.9 (1.5)
  Q2. Hyperglycemia: number analyzed (Participants) | 290 | 286
  Q2. Hyperglycemia | -2.1 (2.1) | -1.6 (2.3)
  Q3. Hypoglycemia: number analyzed (Participants) | 290 | 286
  Q3. Hypoglycemia | 0.1 (1.7) | 0.1 (1.6)
  Q4. Flexibility: number analyzed (Participants) | 290 | 286
  Q4. Flexibility | 0.7 (1.5) | 0.6 (1.5)
  Q5. Convenience: number analyzed (Participants) | 289 | 286
  Q5. Convenience | 0.7 (1.5) | 0.6 (1.5)
  Q6. Understanding of diabetes: number analyzed (Participants) | 290 | 284
  Q6. Understanding of diabetes | 0.6 (1.4) | 0.5 (1.3)
  Q7. Recommend treatment to others: number analyzed (Participants) | 288 | 286
  Q7. Recommend treatment to others | 0.7 (1.5) | 0.7 (1.4)
  Q8. Willingness to continue: number analyzed (Participants) | 290 | 285
  Q8. Willingness to continue | 1.0 (1.8) | 0.9 (1.8)
  Treatment satisfaction summary score: number analyzed (Participants) | 290 | 286
  Treatment satisfaction summary score | 4.6 (7.0) | 4.2 (6.6)

27. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAE)
Description: A TEAE was defined as an adverse event with onset date (or increase in severity) during the on-treatment observation period. The on-treatment observation period represents the time period where subjects were considered exposed to trial product.
Time Frame: Week 0 to week 35
Population: Safety analysis set (SAS) included all subjects exposed to at least one dose of trial product. Number analyzed = number of participants with available data.
Measure: Number; unit: Events
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 289 | 287
Events | 758 | 691

28. Secondary Outcome: Number of Treatment-emergent Severe or Blood Glucose Confirmed Symptomatic Hypoglycaemic Episodes
Description: Hypoglycaemic episodes were defined as treatment emergent if the onset of the episode occurred within the on-treatment observation period, where the subjects were exposed to the trial product. Severe or BG-confirmed symptomatic hypoglycaemia: an episode that was severe according to the ADA classification or blood glucose confirmed by a plasma glucose value below 3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: Week 0 to week 35
Population: as for outcome 27
Measure: Number; unit: Episodes of hypoglycaemia
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 289 | 287
Episodes of hypoglycaemia | 8 | 8

29. Secondary Outcome: Treatment-emergent Severe or Blood Glucose Confirmed Symptomatic Hypoglycaemia Episodes
Description: Number of subjects with treatment-emergent severe or blood glucose confirmed symptomatic hypoglycaemia episodes is presented. Hypoglycaemic episodes were defined as treatment emergent if the onset of the episode occurred within the on-treatment observation period, where the subjects were exposed to the trial product. Severe or BG-confirmed symptomatic hypoglycaemia: an episode that was severe according to the ADA classification or blood glucose confirmed by a plasma glucose value below 3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia.
Time Frame: Week 0 to week 35
Population: as for outcome 27
Measure: Number; unit: Participants
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 289 | 287
Participants | 5 | 7

30. Secondary Outcome: Change in Haematology - Haemoglobin
Description: Mean change from baseline (week 0) to week 30 in haemoglobin. Results are based on the on-treatment observation period where subjects were considered exposed to trial product.
Time Frame: Week 0, week 30
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mmol/L
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 289 | 287
mmol/L | 1.0 (16.0) | 1.0 (0.0)

31. Secondary Outcome: Change in Haematology - Haematocrit
Description: Mean change from baseline (week 0) to week 30 in haematology laboratory parameter haematocrit. Haematocrit is the volume of red blood cells in the total blood. Results are based on the on-treatment observation period where subjects were considered exposed to trial product.
Time Frame: Week 0, week 30
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent change
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 289 | 287
percent change | 1.5 (111.7) | 1.1 (130.9)

32. Secondary Outcome: Change in Haematology - Thrombocytes and Leukocytes
Description: Mean change from baseline (week 0) to week 30 in haematology laboratory parameters thrombocytes and leukocytes. Results are based on the on-treatment observation period where subjects were considered exposed to trial product.
Time Frame: Week 0, week 30
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 10^9 cells/L
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 289 | 287
10^9 cells/L
  Thrombocytes: number analyzed (Participants) | 233 | 245
  Thrombocytes | 18.4 (126.0) | 21.5 (138.9)
  Leukocytes | 0.14 (133.2) | 0.14 (117.3)

33. Secondary Outcome: Change in Haematology - Erythrocytes
Description: Mean change from baseline (week 0) to week 30 in haematology laboratory parameter erythrocytes. Results are based on the on-treatment observation period where subjects were considered exposed to trial product.
Time Frame: Week 0, week 30
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 10^12 cells/L
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 289 | 287
10^12 cells/L | 0.14 (133.2) | 0.14 (117.3)

34. Secondary Outcome: Change in Biochemistry - Calcium, Pottassium and Sodium
Description: Mean change from baseline (week 0) to week 30 in biochemistry laboratory parameters calcium, pottassium and sodium. Results are based on the on-treatment observation period where subjects were considered exposed to trial product.
Time Frame: Week 0, week 30
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mmol/L
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 289 | 287
mmol/L
  Calcium: number analyzed (Participants) | 247 | 260
  Calcium | 0.07 (107.0) | 0.07 (103.8)
  Pottassium: number analyzed (Participants) | 246 | 260
  Pottassium | 0.3 (96.0) | 0.3 (77.3)
  Sodium: number analyzed (Participants) | 247 | 260
  Sodium | 1.8 (65.3) | 1.7 (61.4)

35. Secondary Outcome: Change in Biochemistry - Alkaline Phosphatase, Alanine Aminotransferase and Aspartate Aminotransferase.
Description: Mean change from baseline (week 0) to week 30 in biochemistry laboratory parameters alkaline phosphatase, alanine aminotransferase and aspartate aminotransferase. Results are based on the on-treatment observation period where subjects were considered exposed to trial product.
Time Frame: Week 0, week 30
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mmol/L
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 289 | 287
mmol/L
  Alkaline phosphatase: number analyzed (Participants) | 247 | 260
  Alkaline phosphatase | 5.5 (117.5) | 6.4 (121.0)
  Alanine Aminotransferase: number analyzed (Participants) | 245 | 259
  Alanine Aminotransferase | 5.3 (126.1) | 5.0 (137.7)
  Aspartate Aminotransferase: number analyzed (Participants) | 245 | 257
  Aspartate Aminotransferase | 3.5 (129.9) | 3.1 (119.5)

36. Secondary Outcome: Change in Biochemistry - Amylase and Lipase
Description: Mean change from baseline (week 0) to week 30 in biochemistry laboratory parameters amylase and lypase. Observed data with multiple imputation for missing data is presented. Missing data were imputed using observed data from subjects within the same group defined by actual treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates. Results are based on the on-treatment observation period where subjects were considered exposed to trial product.
Time Frame: Week 0, week 30
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: U/L
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 289 | 287
U/L
  Amylase | 10.3 (124.7) | 8.4 (138.2)
  Lipase | 15.8 (154.6) | 14.0 (154.5)

37. Secondary Outcome: Change in Biochemistry - Creatinine and Bilirubin
Description: Mean change from baseline (week 0) to week 30 in biochemistry laboratory parameters creatinine and bilirubin. Results are based on the on-treatment observation period where subjects were considered exposed to trial product.
Time Frame: Week 0, week 30
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: umol/L
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 289 | 287
umol/L
  Creatinine: number analyzed (Participants) | 247 | 260
  Creatinine | 4.1 (150.2) | 3.6 (150.0)
  Bilirubin: number analyzed (Participants) | 245 | 259
  Bilirubin | 1.9 (167.5) | 2.0 (126.2)

38. Secondary Outcome: Change in Biochemistry - Albumin
Description: Mean change from baseline (week 0) to week 30 in biochemistry laboratory parameter albumin. Results are based on the on-treatment observation period where subjects were considered exposed to trial product.
Time Frame: Week 0, week 30
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: g/dL
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 289 | 287
g/dL | 0.2 (56.8) | 0.2 (55.5)

39. Secondary Outcome: Change in Biochemistry - Estimated Glomerular Filtration Rate (eGFR).
Description: Mean change from baseline (week 0) to week 30 in biochemistry laboratory parameter eGFR. eGFR is calculated using the equation from the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) as defined in KDIGO guidelines. Results are based on the on-treatment observation period where subjects were considered exposed to trial product.
Time Frame: Week 0, week 30
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min/1.73m2
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 289 | 287
mL/min/1.73m2 | 4.0 (97.7) | 4.1 (113.9)

40. Secondary Outcome: Change in Calcitonin
Description: Mean change from baseline (week 0) to week 30 in calcitonin. Results are based on the on-treatment observation period where subjects were considered exposed to trial product.
Time Frame: Week 0, week 30
Population: as for outcome 27
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/L
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 289 | 287
ng/L | 1.3 (165.5) | 1.1 (89.7)

41. Secondary Outcome: Change in Pulse Rate
Description: Mean change from baseline (week 0) to week 30 in pulse rate. Pulse rate is measured as number of heart beats per minute. Results are based on the on-treatment observation period where subjects were considered exposed to trial product. Missing data were imputed using observed data from subjects within the same group defined by randomised treatment, using a regression model including stratification factor as categorical effect and data from baseline and all previous visits as covariates.
Time Frame: Week 0, week 30
Population: Safety analysis set (SAS) included all subjects exposed to at least one dose of trial product.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: beats/min
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
Number analyzed (Participants) | 289 | 287
beats/min | 2.4 (10.1) | 3.9 (10.0)

ADVERSE EVENTS:
Time Frame: From the date of first dose of trial product (week 0) to end of treatment (week 30) + post treatment follow-up of 42 days.
Description: Evaluation of safety was based on safety analysis set (SAS) which comprised of all randomised subjects who received at least one dose of trial product.
  AEs with onset during the on-treatment observation period (the period when subjects were exposed to trial product) were considered treatment-emergent.
Arm/Group | Semaglutide 1.0 mg | Liraglutide 1.2 mg
All-Cause Mortality (participants affected / at risk) | 0/289 | 0/287
Serious Adverse Events (participants affected / at risk) | 17/289 | 22/287
Other Adverse Events (participants affected / at risk) | 139/289 | 113/287
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 1.0 mg (N=289) | Liraglutide 1.2 mg (N=287)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular examination (Investigations) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 2 (2) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 1.0 mg (N=289) | Liraglutide 1.2 mg (N=287)
Abdominal pain (Gastrointestinal disorders) | 15 (18) | 6 (6)
Constipation (Gastrointestinal disorders) | 17 (17) | 10 (13)
Decreased appetite (Metabolism and nutrition disorders) | 30 (31) | 17 (18)
Diarrhoea (Gastrointestinal disorders) | 45 (56) | 35 (43)
Headache (Nervous system disorders) | 27 (37) | 19 (32)
Influenza (Infections and infestations) | 9 (12) | 15 (16)
Nasopharyngitis (Infections and infestations) | 27 (30) | 30 (32)
Nausea (Gastrointestinal disorders) | 62 (88) | 45 (54)
Vomiting (Gastrointestinal disorders) | 29 (43) | 23 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-05-27): https://cdn.clinicaltrials.gov/large-docs/96/NCT03191396/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-27): https://cdn.clinicaltrials.gov/large-docs/96/NCT03191396/SAP_001.pdf